CLINICAL TRIAL: NCT01430689
Title: Prospective, Randomized, Controlled, Observer-Blind Trial to Measure the Efficacy, Safety and Immunogenicity of Trivalent Inactivated Influenza Vaccine and the Safety and Immunogenicity of Quadrivalent Meningococcal Polysaccharide Diphtheria Conjugate Vaccine in Pregnant Malian Women and Their Infants up to 6 Months of Age
Brief Title: Maternal Flu Vaccine Trial in Bamako, Mali
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Milagritos Tapia, Faculty, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00049582
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Influenza
Keywords: Influenza; Pregnancy; Neonates
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inactivated Influenza Vaccine Trivalent Types A and B (Experimental): Women will be vaccinated with Influenza vaccine: Inactivated Influenza Vaccine Trivalent Types A and B
  Interventions: Biological: Inactivated Influenza Vaccine Trivalent Types A and B
- Meningococcal Polysaccharide-Diphtheria Toxoid Conjugate (Active Comparator): Women will be vaccinated with IM injection of Meningococcal Polysaccharide-Diphtheria Toxoid Conjugate Vaccine
  Interventions: Biological: Meningococcal Polysaccharide-Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Inactivated Influenza Vaccine Trivalent Types A and B — Pregnant Woman: Randomization to receive IM injection of Vaxigrip Influenza Vaccine once
  Household and Woman/Infant surveillance
  * Home visits weekly until the infant is born and reaches 6 months of age
  * If the woman, her infant or other household contact has signs and symptoms consistent with Influenza Like Illness (ILI)a nasal and oropharyngeal swab will be obtained
  Other Names: Vaxigrip
  Arms: Inactivated Influenza Vaccine Trivalent Types A and B
Biological: Meningococcal Polysaccharide-Diphtheria Toxoid Conjugate Vaccine — Pregnant Women - Randomized to receive IM injection of Menactra once
  Household and Woman/Infant surveillance
  * Home visits weekly until the infant is born and reaches 6 months of age
  * If the woman, her infant or other household contact has signs and symptoms consistent with Influenza Like Illness (ILI)a nasal and oropharyngeal swab will be obtained
  Other Names: Menactra - Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine; Product No. 49281-589-05
  Arms: Meningococcal Polysaccharide-Diphtheria Toxoid Conjugate

SUMMARY:
The Center for Vaccine Development - Mali is interested in learning if vaccinating a pregnant woman against influenza will protect her infant against this disease. The investigators know that influenza infection, the "flu", affects pregnant women and their infants in Mali. The illness known as flu is caused by a germ (virus) that is passed easily among people. The flu causes symptoms such as fever, cough, sore throat, runny nose, and body aches. Certain groups of people, such as pregnant women and infants, are at risk for having severe disease when they get the flu. Vaccination against influenza is not routinely available to pregnant women in Mali although it is recommended.

Women who wish to participate will have 5 visits to the clinic and weekly visits to the home to follow the health of the woman and her infant when it is born. The investigators will also ask permission to make weekly visits to all children under 5 years of age to follow their health as it relates to influenza infection.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled observer-blind trial measuring the efficacy, safety and immunogenicity of TIV and the safety and immunogenicity of MCV in pregnant women and their infants up to 6 months of age. Women will be recruited in the 3rd trimester of pregnancy and vaccinated with either TIV or MCV. Safety assessments of the women will be completed 30 minutes and 1 week after vaccination, at delivery and 3 and 6 months after delivery. Safety assessments of the infants will be completed at birth and at 3 and 6 months of age. Immunogenicity assessments will include blood sampling of women immediately prior to vaccination, 4 weeks post-vaccination, at delivery and 3 and 6 months after delivery; infants will have cord blood collected at birth and peripheral blood collections at 3 and 6 months of age. Visits to ascertain the costs related to ILI and LCI will also be conducted. The majority of activities conducted in this trial are related to efficacy assessments which will continue until the newborn infant is 6 months of age. We will be conducting case detection for LCI via weekly household visits. In addition, hospital-based surveillance for meningococcal disease will be conducted to measure the efficacy of MCV.

ELIGIBILITY:
Inclusion Criteria:

1. Women in third trimester of pregnancy (≥ 28 weeks gestational age based upon last menstrual period, ultrasound or uterine height).
2. Subject is able to understand and comply with planned study procedures.
3. Subject has provided written informed consent prior to initiation of any study procedures.
4. Subject intends to reside in the study area until her newborn infant is 6 months of age.

Exclusion Criteria:

1. Member of a household which already has a woman who is participating or has participated in this study
2. History of severe reactions following previous immunization with influenza or meningococcal vaccines
3. History of Guillain-Barré Syndrome
4. Known allergy or hypersensitivity to eggs, egg proteins, latex, diphtheria toxoid, or any other components of Vaxigrip and Menactra
5. Known chronic medical condition that in the judgment of the investigator could compromise the evaluation of the study vaccine or puts the subject at risk
6. Known active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
7. Any of the following complications with the ongoing pregnancy: preterm labor (with cervical change), placental abruption, premature rupture of membranes, known major congenital anomaly, or preeclampsia.
8. Acute illness and/or an oral temperature greater than or equal to 37.8 degrees C, within 72 hours of vaccination (This may result in a temporary delay of vaccination)
9. Receipt of any other vaccine, excluding tetanus toxoid, within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines and meningococcal A conjugate vaccine (MenAfriVac)) prior to vaccination in this study
10. Woman who intends to travel out of the study area for the 40 days after delivery
11. Receipt of immunoglobulins and/or any blood products within 30 days prior to the administration of study vaccines
12. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying agents within 90 days prior to administration of study vaccines (including systemic corticosteroids, e.g. prednisone or equivalent > 0.5 mg/kg/day; topical and inhaled steroids are allowed)
13. Any condition which in the opinion of the investigator might compromise the well-being of the participant or compliance with study procedures or interfere with the evaluation of the study vaccines

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4193 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of infants with influenza whose mothers received vaccine at any time during the 3rd trimester | 2 years
  To compare the incidence of laboratory-confirmed influenza (LCI) among infants up to 6 months of age born to mothers immunized with trivalent influenza vaccine (TIV) during the 3rd trimester of pregnancy versus infants born to mothers who received meningococcal conjugate vaccine (MCV) during the 3rd trimester of pregnancy (intention-to-treat (ITT) comparison)

SECONDARY OUTCOMES:
Number of infants with influenza whose mothers received vaccine at least 14 days prior to delivery | 2 years
  To compare the incidence of Laboratory Confirmed Influenza among infants up to 6 months of age born to mothers immunized with TIV during the 3rd trimester of pregnancy versus infants born to mothers who received MCV during the 3rd trimester of pregnancy, for infants born to women immunized ≥ 14 days prior to delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Milagritos D Tapia, MD, Principal Investigator — University of Maryland, College Park; Myron M Levine, MD, DTPH, Study Director — University of Maryland, College Park; Samba O Sow, MD, Principal Investigator — Centre pour le Developpement des Vaccins - Mali
Locations (1):
- Centre pour le Developpement des Vaccins - Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amin AB, Nunes MC, Tapia MD, Madhi SA, Cutland CL, Wairagkar N, Omer SB; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Immunogenicity of influenza vaccines administered to pregnant women in randomized clinical trials in Mali and South Africa. Vaccine. 2020 Sep 22;38(41):6478-6483. doi: 10.1016/j.vaccine.2020.07.020. Epub 2020 Aug 29. PMID 32868130
- [Derived] Omer SB, Clark DR, Madhi SA, Tapia MD, Nunes MC, Cutland CL, Simoes EAF, Aqil AR, Katz J, Tielsch JM, Steinhoff MC, Wairagkar N; BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Efficacy, duration of protection, birth outcomes, and infant growth associated with influenza vaccination in pregnancy: a pooled analysis of three randomised controlled trials. Lancet Respir Med. 2020 Jun;8(6):597-608. doi: 10.1016/S2213-2600(19)30479-5. PMID 32526188
- [Derived] Clark DR, Omer SB, Tapia MD, Nunes MC, Cutland CL, Tielsch JM, Wairagkar N, Madhi SA; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Influenza or Meningococcal Immunization During Pregnancy and Mortality in Women and Infants: A Pooled Analysis of Randomized Controlled Trials. Pediatr Infect Dis J. 2020 Jul;39(7):641-644. doi: 10.1097/INF.0000000000002629. PMID 32379201
- [Derived] Omer SB, Clark DR, Aqil AR, Tapia MD, Nunes MC, Kozuki N, Steinhoff MC, Madhi SA, Wairagkar N; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Maternal Influenza Immunization and Prevention of Severe Clinical Pneumonia in Young Infants: Analysis of Randomized Controlled Trials Conducted in Nepal, Mali and South Africa. Pediatr Infect Dis J. 2018 May;37(5):436-440. doi: 10.1097/INF.0000000000001914. PMID 29443825
- [Derived] Tapia MD, Sow SO, Tamboura B, Teguete I, Pasetti MF, Kodio M, Onwuchekwa U, Tennant SM, Blackwelder WC, Coulibaly F, Traore A, Keita AM, Haidara FC, Diallo F, Doumbia M, Sanogo D, DeMatt E, Schluterman NH, Buchwald A, Kotloff KL, Chen WH, Orenstein EW, Orenstein LAV, Villanueva J, Bresee J, Treanor J, Levine MM. Maternal immunisation with trivalent inactivated influenza vaccine for prevention of influenza in infants in Mali: a prospective, active-controlled, observer-blind, randomised phase 4 trial. Lancet Infect Dis. 2016 Sep;16(9):1026-1035. doi: 10.1016/S1473-3099(16)30054-8. Epub 2016 May 31. PMID 27261067